CLINICAL TRIAL: NCT02195947
Title: Does the Addition of Growth Hormone to the Invitro Fertilization/ Intracytoplasmic Sperm Injection Antagonist Protocol Improve Outcome in Poor Responders? A Randomized Controlled Trial
Brief Title: Antagonist Protocol in Poor Responders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Ahmed Bassiouny, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 72014
Record Dates: First submitted 2014-07-18; First posted 2014-07-21 (Estimated); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Female Infertility Due to Diminished Ovarian Reserve
Keywords: Growth hormone; IVF/ICSI; Poor responder; Antagonist protocol
MeSH Terms: interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antagonist and Growth hormone (Experimental): HMG IM daily was administrated from day 2 of the cycle. The GnRH antagonist (Cetrotide, Serono, Geneva, Switzerland) was given when the leading follicle was from 12 to 14 mm, at a daily dose of 0.25 mg SC. Growth hormone (Norditropin, Novo nordisk) was administrated on day 6 of HMG stimulation daily in a dose of 2.5 mg S.C. till the day of hCG administration.
  Interventions: Drug: Growth Hormone
- Antagonist (No Intervention): HMG IM daily was administrated from day 2 of the cycle. The GnRH antagonist (Cetrotide, Serono, Geneva, Switzerland) was given when the leading follicle was from 12 to 14 mm, at a daily dose of 0.25 mg SC

INTERVENTIONS:
Drug: Growth Hormone — Growth hormone (Norditropin, Novo nordisk) was administrated on day 6 of HMG stimulation daily in a dose of 2.5 mg S.C. till the day of hCG administration.
  Other Names: Norditropin, Novo nordisk
  Arms: Antagonist and Growth hormone

SUMMARY:
The effect of use of the growth hormone with antagonist protocol on the outcome of the IVF/ICSI cycles in poor responders.

DETAILED DESCRIPTION:
Two groups of poor responder female patients planned to receive the antagonist IVF/ICSI protocol are randomized to whether or not to add growth hormone to their protocol.

ELIGIBILITY:
Inclusion Criteria:

* females fulfilling the criteria of the ESHRE consensus 2011:
* at least two of the following three features must be present:
* dvanced maternal age (≥40 years) or any other risk factor for POR
* previous POR (≤3 oocytes with a conventional stimulation protocol)
* an abnormal ovarian reserve test (i.e. AFC ,5-7 follicles or AMH ,0.5 -1.1 ng/ml).

Exclusion Criteria:

* women who suffer from any other cause of infertility other than poor ovarian reserve
* refusal of the patient to consent for using her data in the study.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Live birth rate | Up to 9 months

SECONDARY OUTCOMES:
Clinical pregnancy rate | Up to 5 weeks

OTHER OUTCOMES:
Chemical pregnancy rate | 5 weeks
Early miscarriage rate | Up to 12 weeks
Ongoing pregnancy rate | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yomna A Bayoumi, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr Al Aini, Cairo, Egypt

REFERENCES:
- [Derived] Bassiouny YA, Dakhly DMR, Bayoumi YA, Hashish NM. Does the addition of growth hormone to the in vitro fertilization/intracytoplasmic sperm injection antagonist protocol improve outcomes in poor responders? A randomized, controlled trial. Fertil Steril. 2016 Mar;105(3):697-702. doi: 10.1016/j.fertnstert.2015.11.026. Epub 2015 Dec 13. PMID 26690008